CLINICAL TRIAL: NCT03870048
Title: Transcranial Direct Current Stimulation to Lower Neuropathic Pain and Fatigue in People With Multiple Sclerosis
Brief Title: tDCS to Lower Neuropathic Pain and Fatigue in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: jkamholz (Unknown); Workman, Craig D., PhD (Individual)
Responsible Party: Principal Investigator, Thorsten Rudroff, Principal Investigator, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201812729
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All Study Participants/tDCS or SHAM (Experimental): tDCS Block: The participant will receive tDCS for 20 min at an intensity of 2 mA while seated comfortably and quietly in a room. The intensity will start at 0 mA and will be incrementally increased to 2mA over the initial 30 seconds. At the 19:30 minute time point, the current will gradually be reduced from 2 mA to 0 mA.
  Sham block: Identical to the tDCS block, except the participants will only receive the initial 30 seconds of ramp-up, after which the current will be set to 0 for the remainder of the 20 minutes.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.

SUMMARY:
The purpose of this study is to investigate the effects of transcranial direct current stimulation (tDCS) on neuropathic pain and fatigue in people with MS. The investigators will conduct tDCS or sham on 5 consecutive days. They will evaluate pain and fatigue with specific questionnaires and measure fatigability with an isokinetic device.

The research question is whether tDCS can lessen neuropathic pain and increase fatigue resistance in people with MS. It is hypothesized, that less neuropathic pain and increased fatigue resistance after the tDCS sessions.

DETAILED DESCRIPTION:
Prospective participants, men and women with MS, will be recruited. To accomplish this study, 20 participants will need to complete 2 randomly-ordered blocks of protocols (tDCS or sham), separated by at least one week. Each block involves 5 daily sessions at the INPL. The duration of each session will be approximately one hour and will be completed at the same time of day for each subject. The investigators expect data collection to last 6 months. Each session will be a combination of questionnaires, leg strength assessment, and an isokinetic fatigue test.

Leg strength assessment: Isokinetic (concentric/concentric) flexion and extension of the knee at 60°/s will performed five times to determine the more-MS affected leg. When strength difference between the left and right legs is less than 10%, the more affected side will be based on the participant's self-report.

Isokinetic fatigue test: Participant's will perform 40 consecutive repetitions of isokinetic concentric/concentric flexion and extension of the knee on the more-affected leg at 120 degree/sec.

In the initial session (i.e., Block 1, Session 1) subjects will 1) be consented, 2) complete the Patient Determined Disease Steps (PDDS) questionnaire, 3) the Fatigue Severity Scale (FSS), 4) Neuropathic Pain Questionnaire (NPQ), 5) Visual analog scale (VAS), 6) perform a leg strength assessment, 7) perform an isokinetic fatigue test, and 8) undergo either tDCS or sham treatment, depending on the randomized block.

tDCS treatment protocol: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit. The two protocols blocks (tDCS or sham) will be performed in randomized order.

tDCS Block: The participant will receive tDCS for 20 min at an intensity of 2 mA while seated comfortably and quietly in a room. The intensity will start at 0 mA and will be incrementally increased to 2mA over the initial 30 seconds. At the 19:30 minute time point, the current will gradually be reduced from 2 mA to 0 mA.

Sham block: Identical to the tDCS block, except the participants will only receive the initial 30 seconds of ramp-up, after which the current will be set to 0 for the remainder of the 20 minutes.

The remaining sessions of first block (i.e. Block 1, Sessions 2-5) will be as follows: In Sessions 2 and 4, the subjects get the tDCS or sham treatment, after which they will complete the fatigue and pain questionnaires (FSS and NPQ). Sessions 3 will be the same as Sessions 2 and 4, except that the isokinetic fatigue test will be performed at the beginning (i.e., before the tDCS or sham treatment). Session 5 will start with tDCS or sham treatment, then the isokinetic fatigue test, and finally the fatigue and pain questionnaires.

Block 2 will be completed in the same manner as Block 1, except that the subjects will not redo the PDDS, VAS, and BDI in Session 1 and the treatment will shift to either tDCS or sham, depending on how the blocks were randomized.

Duration of Relief - If the participant indicates any reduction in pain following the previous day's tDCS session, they will be asked to estimate how long their pain was reduced following the session. Additionally, one week following the last testing session (i.e., Block 2, Session 5), participants will be contacted via telephone and asked the following questions:

1. Was tDCS effective at reducing the subject's pain?
2. If so, how long did the subject notice a reduction in pain following your final tDCS session?
3. Have the subject reduced his/her use of pain relieving medications since your last tDCS session?

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with Multiple Sclerosis
* 18-70 yrs. of age, moderate disability (Patient Determined Disease Steps (PDDS) core 2-6)
* Self-reported differences in function between legs
* Able to walk for 6 min
* Presenting with chronic, drug-resistant, neuropathic pain.

Exclusion Criteria:

* Relapse within last 60 days
* High risk for cardiovascular disease (ACSM risk classification)
* Changes in disease modifying medications within last 45 days
* Concurrent neurological/neuromuscular disease
* Hospitalization within last 90 days
* Diagnosed depression
* Inability to understand/sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- tDCS Effects on Pain and Fatigue: tDCS Block: The participant will receive tDCS for 20 min at an intensity of 2 mA while seated comfortably and quietly in a room. The intensity will start at 0 mA and will be incrementally increased to 2mA over the initial 30 seconds. At the 19:30 minute time point, the current will gradually be reduced from 2 mA to 0 mA.
  transcranial direct current stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.
Period: SHAM Effects on Pain and Fatigue
Arm/Group | tDCS Effects on Pain and Fatigue
Started | 6
Completed | 6
Not Completed | 0
Period: tDCS Effects on Pain and Fatigue
Arm/Group | tDCS Effects on Pain and Fatigue
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- tDCS Effects on Pain and Fatigue: tDCS Block: The participant will receive tDCS for 20 min at an intensity of 2 mA while seated comfortably and quietly in a room. The intensity will start at 0 mA and will be incrementally increased to 2mA over the initial 30 seconds. At the 19:30 minute time point, the current will gradually be reduced from 2 mA to 0 mA.
  transcranial direct current stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.
  Sham block: Identical to the tDCS block, except the participants will only receive the initial 30 seconds of ramp-up, after which the current will be set to 0 for the remainder of the 20 minutes.
Arm/Group | tDCS Effects on Pain and Fatigue
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.7 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Neuropathic Pain Questionnaire (NPQ) Contains 12 Items.
Description: The participant is asked to use items to rate their pain as it usually feels. They have to indicate a number which represents their pain on each scale. For example, if someone has no burning pain, the person would rate the first item "0". If the person has the worst burning pain imaginable, he/she would rate it "100". If neither of those fits his/her pain because it is in between, the participant has to choose a number which fits his/her pain.
Time Frame: 2 Months
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Sham Effects on Pain and Fatigue: Sham block: Identical to the tDCS block, except the participants will only receive the initial 30 seconds of ramp-up, after which the current will be set to 0 for the remainder of the 20 minutes.
  transcranial direct current stimulation: A tDCS device (Soterix) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The positive electrode will be placed over the motor cortex representation of the more affected leg, and a second electrode will be placed on the forehead above the contralateral orbit.
Arm/Group | tDCS Effects on Pain and Fatigue | Sham Effects on Pain and Fatigue
Number analyzed (Participants) | 6 | 6
Points | 21.3 (19.5) | 10.3 (13.5)

2. Secondary Outcome: Fatigue Severity Scale (FSS) Contains Nine Statements That Attempt to Explore Severity of Fatigue Symptoms.
Description: The FSS questionnaire The participant has to read each statement and circle a number from 1 to 7, depending on how appropriate they felt the statement applied to them over the preceding week. A low value indicates that the statement is not very appropriate whereas a high value indicates agreement (1 disagree, 7 agree).
Time Frame: 2 Months
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | tDCS Effects on Pain and Fatigue | Sham Effects on Pain and Fatigue
Number analyzed (Participants) | 6 | 6
Points | 4 (2) | 6 (1)

ADVERSE EVENTS:
Time Frame: 350 Days
Arm/Group | tDCS Effects on Pain and Fatigue | Sham Effects on Pain and Fatigue
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03870048/Prot_SAP_006.pdf